CLINICAL TRIAL: NCT04587999
Title: Quick-Wee Versus Bladder Stimulation to Collect Midstream Urine From Pre-continent Infants: a Randomized Controlled Trial
Brief Title: Quick-Wee Versus Bladder Stimulation System to Collect Midstream Urine From Pre-continent Infants
Acronym: ES-Stimquick U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-HPNCL-04
Record Dates: First submitted 2020-09-25; First posted 2020-10-14 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bladder stimulation (Experimental)
  Interventions: Other: bladder stimulation
- Quick wee (Active Comparator)
  Interventions: Other: Quick wee

INTERVENTIONS:
Other: bladder stimulation — The bladder stimulation technique requires the presence of 2 people:
  * The child must be held by an adult (caregiver or parent) under the armpits, legs dangling.
  * the first person (the investigator), performs the stimulation technique consisting of: rapid tapping (frequency of about 100 / min), over the pubic area, at the level of the bladder, alternated with external rotational movements of the pits lumbar, in the kidneys. Alternate these 2 maneuvers every 30 seconds.
  * The second person starts the stopwatch at the start of the stimulation, and is about to collect the urine, 2nd jet in a sterile pot
  * The maneuver ends as soon as urine is obtained, and will be stopped after 5 minutes in case of failure.
  Arms: bladder stimulation
Other: Quick wee — The Quick wee technique requires the presence of only one person:
  Stimulation of the suprapubic area by circular movements, with a cold and wet compress held by sterile forceps.
  Collection of urine in a sterile container.
  Arms: Quick wee

SUMMARY:
Urinary tract infections are common in infants. Obtaining urine from pre-continent children can be difficult and time consuming. The method of collection must balance reliability, speed, low rate of contamination, and invasiveness.

According to the American Academy of Pediatrics, midstream clean-catch urine is an acceptable method to diagnose urinary tract infections. However, it is impractical in pre-continent children.

Recently, two quick, safe and effective methods have been reported in the literature:

* The Quick-wee method: it consists in stimulating the suprapubic area with a cold and wet compress to obtain urines.
* The bladder stimulation method : the child is held under the armpits with legs dangling and a physician taps the suprapubic area and massages lumbar area alternatively.

However, advanced age, high weight, and level of discomfort during bladder stimulation were significantly associated with failure to obtain urines.

DETAILED DESCRIPTION:
Urinary tract infections (UTI) are common in infants. The diagnosis of a UTI has important implications for follow-up, and delayed treatment can result in morbidity, including renal scarring and serious bacterial infection.

Obtaining urine from pre-continent children can be difficult and time consuming, the method of collection must balance reliability, speed, low rate of contamination, and invasiveness The actual guidelines recommend suprapubic aspiration or bladder catheterization for collection of urine sample in pre-continent children, but these methods are invasive.

The most common way to collect urines in infants is the use of a sterile collection bag. This is an easy technique, but time consuming and responsible for high rate of contamination, leading to false positives.

According to the American Academy of Pediatrics, midstream clean-catch urine is an acceptable method to diagnose urinary tract infection. However, it is impractical in pre-continent children.

Recently, two quick, safe and effective methods have been reported in the literature:

* The Quick-wee method: it consists in stimulating the suprapubic area with a cold and wet compress to obtain urines.
* The bladder stimulation method: the child is held under the armpits with legs dangling and a physician taps the suprapubic area and massages lumbar area alternatively.

However, advanced age, high weight, and level of discomfort during bladder stimulation were significantly associated with failure to obtain urines.

Futhermore, even if urine collection in pre-continent children most often concerns urinary tract infections, these techniques could also be used to look for a metabolic abnormality, an uropathy or a nephropathy (urine electrolyte concentrations, proteinuria, hematuria).

The aim of the study is to compare the effectiveness of two non-invasive midstream urine collection methods in pre-continent children : "the Quick-Wee method" and "the Bladder stimulation method".

The investigators will also compare in the two groups the time required to obtain urine sample, the comfort of the infant during urine collection and the quality of urines.

Finally, for each technique will be analyzed the risk factors associated with failure in obtaining urine sample

ELIGIBILITY:
Inclusion Criteria:

* Infants under the age of 1 year, pre-continent, before walking
* For whom an urine sample is required for the diagnosis of a urinary tract infection, uropathy, nephropathy, metabolic disease
* Obtaining the authorization by one of the two parents or the holder of parental authority
* Affiliation to a national social security scheme

Exclusion Criteria:

* Do exhibiting signs of vital distress
* Withdrawal of informed consent by parents or holders of parental authority
* External genitalia or urinary tract malformation
* Bladder dysfunction

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
volume of urine collection to measure the effectiveness of two techniques | at the end of intervention completion, an average 30 minutes
  measure of success of the urine collection technique is determined by collecting at least 2 millimeters of urine in less than 5 minutes

SECONDARY OUTCOMES:
time needed to obtain urines | at the end of intervention completion, an average 30 minutes
  measure of times needed to obtain urines in minutes and seconds
patient comfort | through intervention completion, an average 30 minutes
  pain is measured by Evaluation ENfant DOuLeur (EVENDOL) scale while the technique is performed. EVENDOL is a pain scale for children under 7. A pain scale validated for children from birth to 7 years. Score ranges from 0 to 15.
  Treatment threshold: 4/15.
Bacterial contamination rates of urine samples | at 48 hours after inclusion
  Measure of bacterial contamination of urine sample is by:
  * numeration the growth of two or more micro-organisms,
  * Or numeration the presence of a non-uropathogenic germ (lactobacilli, Staphylococcus Coagulase negative, Corynebacterium),
  * or numeration a bacteriuria> 0 colony forming unit(CFU)/millimeters (mL) but <10˄4 CFU / ml for bladder catheterization and <10˄5 CFU / mL for clean catch urine collected by bladder stimulation, or leukocyturia <10˄4 / mL
collection of patient data to define risk factors associated with the failure of the bladder stimulation techniques | through intervention completion, an average 30 minutes
  collection patient data : pain, weight, sex, age, last food and time since last collect urine The goal is to define potential risk factors to failure urine collection (urinary sample quantity < 2 millimeters or no urinary sample collected)

CONTACTS AND LOCATIONS:
Locations (3):
- Centre Hospitalier Universitaire de Sainte-Justine, Montreal, Canada
- France (2):
  - Centre Hospitalier Antibes Juan les Pins, Antibes
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice

REFERENCES:
- [Derived] Marchal S, Janicot J, Salicis J, Demonchy D, Herisse AL, Olla M, Rancurel A, Haas H, Berard E, Breaud J, Bernardor J, Ribet C, Freyssinet E, Donzeau D, Desmontils J, Schori-Fortier C, Fontas E, Tran A. Quick-Wee versus bladder stimulation to collect midstream urine from precontinent infants under 1 year of age: a study protocol for a randomised controlled trial (ES.Stimquick.U). BMJ Open. 2021 Sep 16;11(9):e046324. doi: 10.1136/bmjopen-2020-046324. PMID 34531206